CLINICAL TRIAL: NCT06194682
Title: "Valutazione Dell'Epidemiologia e Dei Risultati Clinici Nel Trattamento Artroscopico Delle Lesioni Del Legamento Crociato Anteriore"
Brief Title: Anterior Cruciate Ligament Study
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: ACL(L2104)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: ACL Injury; ACL; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction — Anterior cruciate ligament arthroscopic reconstruction

SUMMARY:
This retrospective, prospective observational study aims to evaluate the epidemiology and rate of anterior cruciate ligament re- rupture after surgery in patients treated from January 2020 to December 2030 by recording both clinically and radiographically ligament reconstruction.

The primary outcome is the rate of rupture of the anterior cruciate ligament as measured by the Lachmann test in which a positive value for re-rupture is an anterior translation of the tibia greater than 10mm relative to the femur Secondary Objectives: Verify predisposing factors to anterior cruciate ligament injuries (so anatomical factors such as tibial slope, trochlear groove), demographic factors (age, sex, weight, sports played), and the rate of return to sports, quality of life via questionnaires, and arthrosis at the operated knee

ELIGIBILITY:
Inclusion Criteria:

* - Males and females- attained skeletal maturity
* 18-65 inclusive
* Patients operated on anterior cruciate ligament reconstruction surgery at the Hospital's Casco unit from 2010 to 2030
* Signature informed consent for patients who will be operated on in the prospective phase (from CE approval date to 2030)

Exclusion Criteria:

* failure to reach skeletal maturity

  * Concomitant ligamentous injuries (pcl, mcl, lcl)
  * Neuropsychiatric illness, developmental disorders
  * Pregnant women through self-declaration or breastfeeding
  * Minors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone and will undergo anterior cruciate ligament reconstruction surgery at the CASCO Team between January 2020 and December 2030. Clinical data, any questionnaires, scores, and radiographic parameters were collected at the same time as the visits and prescribed procedures according to the clinical routine of the department. No additional services will be prescribed by virtue of participation in this study
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Rerupture rate | 10 years
  rate of rerupture rare evaluated with anterior tibial translation

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided